CLINICAL TRIAL: NCT03320265
Title: Double-blind, Randomised, Placebo-controlled, Multicentre, Phase IIa Study to Investigate the Effect of PC-mAb on Arterial Inflammation in Subjects With Elevated Lipoprotein a
Brief Title: Phosphorylcholine PC-mAb Effects in Subjects With Elevated Lipoprotein a
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated
Sponsor: Athera Biotechnologies AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATH3G10-005
Record Dates: First submitted 2017-10-10; First posted 2017-10-25 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Arterial Inflammation; Cardiovascular Diseases
Keywords: Phosphorylcholine human monoclonal antibody; Lipoprotein a
MeSH Terms: conditions — Arteritis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC-mAb (Experimental): Phosphorylcholine human monoclonal antibody, i.v. infusions
  Interventions: Drug: PC-mAb
- Placebo (Placebo Comparator): Placebo to PC-mAb, i.v. infusions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PC-mAb — Monthly treatment for 3 months (4 administrations)
  Arms: PC-mAb
Drug: Placebo — Monthly treatment for 3 months (4 administrations)
  Arms: Placebo

SUMMARY:
Inflammation and abnormal amount of lipids in the blood are key factors for the development and progression of atherosclerosis (thickening of the artery wall) and cardiovascular disease. Lipoprotein (a) is a pro-inflammatory plasma lipoprotein that is believed to be a risk factor for cardiovascular diseases. Vascular inflammation generates a range of effects, including endothelial dysfunction and migration of white blood cells into the vessel wall, which results in increased risk of cardiovascular events.

This study is designed to assess the effects of multiple monthly intravenous infusions with the fully human antibody called PC-mAb, in subjects with elevated lipoprotein (a).

ELIGIBILITY:
Major inclusion criterion:

* Lp(a) above 50 mg/dL at screening

Major exclusion criteria:

* Medical history of myocardial infarction (MI) or stroke within 12 months of screening
* Ongoing or paroxysmal atrial fibrillation
* Clinically overt heart failure
* Hypertension defined as ≥180/100 mmHg
* Diabetes mellitus
* Systemic autoimmune diseases requiring treatment
* Cancer, excluding basal cell carcinoma, within the last five years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Monocyte function | From baseline (Day 1) to visit 11 (Day 85)
  Change in transendothelial migration (TEM) in monocytes isolated from treated subjects

SECONDARY OUTCOMES:
Arterial inflammation | From baseline (Day 1) to visit 11 (Day 85)
  Change in tissue to background ratio (TBRmax) in common carotid arteries by fluorodeoxyglucose-positron emission tomography/computed tomography (FDG-PET/CT)
Arterial stiffness | From baseline (Day 1) to visit 11 (Day 85)
  Change in pulse wave velocity (PWV) (m/sec)
Adverse events (AEs)/serious AEs (SAEs) | From baseline (Day 1) to visit 11 (Day 85)
  Incidence of AEs/SAEs
Vital signs, height | At screening (Day -63 to -1)
  in cm
Vital signs, body weight | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  in kg
Vital signs, blood pressure | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  in mmHg
Vital signs, hear rate | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  in bpm
Vital signs, body temperature | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  in °C
Physical examination including review of all organ systems | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  Any abnormalities will be recorded
Electrocardiogram (ECG), PR (PQ) | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  12-lead ECG; PR (PQ) interval (in msec) will be measured and reported descriptively; any abnormalities will be recorded
ECG, QRS | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  12-lead ECG; QRS interval (in msec) will be measured and reported descriptively; any abnormalities will be recorded
ECG, QT | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  12-lead ECG; QT interval (in msec) will be measured and reported descriptively; any abnormalities will be recorded
ECG, QTcF | At screening (Day -63 to -1), Day 1, Day 28, Day 56, Day 84 and end of study (Day 143)
  12-lead ECG; QTcF interval (in msec) will be measured and reported descriptively; any abnormalities will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Eric SG Stroes, MD, Prof., Principal Investigator — Department of Vascular Medicine, Academic Medical Center, Amsterdam, the Netherlands
Locations (2):
- Department of Vascular Medicine, Academic Medical Center, Amsterdam, Netherlands
- CTC Clinical Trial Consultants AB, Uppsala, Sweden